CLINICAL TRIAL: NCT06709833
Title: Meningioma and Embolism Thrombosis Risk & Investigation of Coagulation
Acronym: 001_2024_BO2
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 001_2024_BO2
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Meningeoma; Thrombembolism; Surgical Resection
Keywords: meningeoma; thrombembolism; tissue-factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Meningioma resection: patients undergoing resection for meningioma
- Glioma resection: Patients undergoing glioma resection as a control cohort for meningioma patients
- Healthy controls: Healthy controls without tumor and surgical resection

SUMMARY:
Despite being generally benign tumors, meningiomas are associated with an increased risk for thrombembolic complications after surgical resection. The molecular mechanisms underlying this circumstance are still unknown.

In this prospective observational trial, the investigators aim to evaluate the changes in coagulation and platelet function caused by tumor resection.

Blood samples are obtained by patients undergoing meningioma resection before and immediately after resection to detect said changes.

As a control cohort, blood samples are obtained from patients undergoing resection for glioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing resection for meningioma or
* Patients undergoing resection for glioma or
* Healthy controls
* written consent for study participation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial tumors
  1. meningeoma
  2. glioma (control)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Tissue factor | duration of surfical tumor resection (a few hours)
  Concentration of tissue factor at pre-surgery and immediately after tumor resection (during close-up).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital for Anaesthesiology and Intensive Care Medicine, Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No